CLINICAL TRIAL: NCT03736460
Title: A Mindfulness-based Intervention for Breast-cancer Patients With Cognitive Impairment After Chemotherapy: Study Protocol of a Three-Group Randomized Controlled Trial
Brief Title: Cancer Related Cognitive Impairment After Chemotherapy: Evaluation of Potential Therapeutic Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Katleen Van der Gucht, Senior Investigator at Leuven Mindfulness Centre | KU Leuven, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S59396
Record Dates: First submitted 2018-11-01; First posted 2018-11-09 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Mindfulness; Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-based intervention (Experimental)
  Interventions: Behavioral: Mindfulness
- Physical training (Active Comparator)
  Interventions: Behavioral: Physical training
- Wait-list (No Intervention)

INTERVENTIONS:
Behavioral: Mindfulness — The mindfulness-based intervention adheres to a standardized protocol developed from the MBSR curriculum (Kabat-Zinn, 1990). The program consists of four 3h group sessions spread over 8 weeks. Each session consists of guided experiential mindfulness exercises (e.g. focus on the breath, body scan, breathing space, mindful movement, sitting meditation), sharing of experiences of these exercises, reflection in small groups, psycho-education (e.g. stress, depression, fear of cancer recurrence, self-care) and review of home practices.
  Arms: Mindfulness-based intervention
Behavioral: Physical training — This intervention is based on the recommended levels of physical activity for adults aged 18 - 64 year from the World Health Organization. These recommendations are the same for women after a breast cancer treatment (Schmitz et al., 2010). Just as the mindfulness intervention this will consist of four 2h group sessions spread over 8 weeks. Each session will consist of psycho-education (e.g. basics of movement, advantages of physical activity, training-principles), endurance and resistance training, stretching, balance and relaxation exercises, sharing of experiences of these exercises and review of home practices.
  Arms: Physical training

SUMMARY:
Background: Mindfulness has been applied to improve after cancer care by enhancing psychological well-being; however, little is known about its impact on cognitive impairment experienced by cancer patients after chemotherapy. Mindfulness may be relevant in tackling cognitive impairment by decreasing emotional distress and fatigue, by decreasing inflammation, and by strengthening brain functional connectivity. The aim of the present study protocol is to evaluate the efficacy and mechanisms of a mindfulness-based intervention to reduce cognitive impairment in breast-cancer patients after chemotherapy.

Methods: The present study is a three-group randomized controlled trial with assessments at baseline, one-three weeks after the intervention and at three months follow-up. One hundred twenty breast cancer patients who ended treatment minimum 6 months and maximum 5 years before and who have cognitive complaints will be enrolled. They will be randomized into one of the following three study arms: (1) a mindfulness-based intervention group (n=40), (2) an active control condition based on physical training (n=40), or (3) a waitlist control group (n=40). Both the mindfulness-based intervention and the active control condition exist of four group sessions (3 hours for the mindfulness condition and 2 hours for the physical training) spread over 8 weeks. The primary outcomes will be cognitive complaints as measured by the cognitive failure questionnaire and changes in brain functional connectivity in the attention network. Secondary outcomes will be (1) levels of emotional distress, fatigue, mindfulness; (2) neurocognitive tests; (3) structural and functional brain changes using MR imaging, and (4) inflammation.

Discussion: The study will examine the impact of a mindfulness-based intervention on cognitive impairment in breast-cancer patients. If the findings of this study confirm the effectiveness of a mindfulness-based program to reduce cognitive impairment, it will be possible to improve quality of life for ex-cancer patients. We will inform health care providers about the potential use of a mindfulness-based intervention as a non-pharmaceutical, low-threshold mental health intervention to improve cognitive impairment after cancer.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of breast cancer at an early stage with or without solitary metastases (except solitary brain metastases)
* completed treatment (surgery and chemotherapy) minimum 6 months and maximum 5 years before
* significant cognitive complaints as measured by the Cognitive Failure questionnaire (CFQ total score > mean study Ponds + 1 SD or on 2 or more of the CFQ extra questions (T/E) > mean study Ponds + 1 SD; (Ponds, Van Boxtel, & Jolles, 2006))
* have sufficient understanding of Dutch

Exclusion Criteria:

* a history of mental retardation, psychiatric and or neurological disorder
* previous participation in a mindfulness training

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Subjective cognitive function | Measurements will take place at baseline (i.e. one to three weeks before randomization), one to three weeks after the intervention and three months after the intervention.
  Change in scores on the Cognitive failure questionnaire
Changes in brain functional connectivity in the attention network | Measurements will take place at baseline (i.e. one to three weeks before randomization), one to three weeks after the intervention and three months after the intervention.
  fMRI imaging

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Deprez, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Van der Gucht K, Melis M, Ahmadoun S, Gebruers A, Smeets A, Vandenbulcke M, Wildiers H, Neven P, Kuppens P, Raes F, Sunaert S, Deprez S. A mindfulness-based intervention for breast cancer patients with cognitive impairment after chemotherapy: study protocol of a three-group randomized controlled trial. Trials. 2020 Mar 23;21(1):290. doi: 10.1186/s13063-020-4204-8. PMID 32293533